CLINICAL TRIAL: NCT01623544
Title: A U.S. Retrospective Database Analysis Evaluating the Comparative Effectiveness of Budesonide/Formoterol Combination (BFC) and Fluticasone Propionate/Salmeterol Combination (FSC) Among Asthma Patients
Brief Title: Asthma Comparative Effectiveness Study
Acronym: Asthma CER
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: RWE-000015
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Asthma
Keywords: Asthma; Comparative Effectiveness; Symbicort
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Symbicort: BFC patients new to ICS/LABA combination therapy
- Advair: FSC patients new to ICS/LABA combination therapy

SUMMARY:
The objective of this study is to compare the real-world effectiveness of BFC and FSC in asthma patients new to ICS/LABA combination therapy in a population of U.S. health plan enrollees.

DETAILED DESCRIPTION:
A U.S. retrospective database analysis evaluating the comparative effectiveness of budesonide/formoterol and fluticasone propionate/salmeterol among asthma patients

ELIGIBILITY:
Inclusion Criteria:

* Continuous health plan enrollment for 12 months before and after index Rx
* At least two prescription fills for BFC or FSC within 12 months
* Asthma claims diagnosis, and 12 to 64 years of age at the time of first prescription

Exclusion Criteria:

* Evidence of COPD
* Claims diagnosis of any of inflammatory diseases or cancer
* Presence of Rx for more than one type of ICS/LABA combination on index date
* Chronic steroid use or Xolair use prior to ICS/LABA index treatment

Ages: 12 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Health plan members with asthma aged 12 to 64 years receiving two or more prescriptions for BFC or FSC during 6/1/2007-9/30/2010 who are naive to ICS/LABA combination therapy.
Sampling Method: Non-Probability Sample
Enrollment: 6086 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Rate of asthma exacerbations | 12 months
  The rate is defined as the total number of asthma exacerbations for all patients in the cohort divided by the total number of person years. An asthma exacerbation is defined as any of three conditions: Asthma related inpatient hospitalization or Asthma related emergency department visit or Oral corticosteroid use.
Asthma Related Inpatient Hospitalizations | 12 months
Asthma Related Emergency Department visits | 12 months
Use of Oral Corticosteroids (OCS) | 12 months
  A pharmacy claim for any of the OCS medications

SECONDARY OUTCOMES:
Asthma controller medication use (SABA, ICS, LABA, LTRA, XOLAIR, THEOPHYLLINE) | 12 months
  Asthma controller use (0 vs. 1 and total number of fills for each).
Asthma Related Healthcare Utilization | 12 months
  Asthma Related Healthcare Utilization: Outpatient/office visits, Inpatient length of stay, ICU admission and length of stay.
Asthma Related Healthcare costs | 12 months
  Asthma Related Healthcare costs (plan paid, patient paid and plan + patient paid)costs of all Asthma related medication and Asthma related outpatient/office, ED and Inpatient visits.

REFERENCES:
- [Derived] Tunceli O, Williams SA, Kern DM, Elhefni H, Pethick N, Wessman C, Zhou S, Trudo F. Comparative effectiveness of budesonide-formoterol combination and fluticasone-salmeterol combination for asthma management: a United States retrospective database analysis. J Allergy Clin Immunol Pract. 2014 Nov-Dec;2(6):719-26. doi: 10.1016/j.jaip.2014.07.016. Epub 2014 Oct 3. PMID 25439363